CLINICAL TRIAL: NCT03949036
Title: Comparison of Two Different Preload Targets of Stroke Volume Variation During Kidney Transplantation: A Randomized Controlled Trial
Brief Title: Comparison of Two Different Preload Targets of Stroke Volume Variation During Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Won Ho Kim, MD, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1811-028-983
Record Dates: First submitted 2019-05-11; First posted 2019-05-14 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Kidney Transplant; Complications; Renal Failure Chronic
Keywords: kidney transplantation; preload index; stroke volume variation; goad-directed therapy
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial of two parallel groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients do not know which group they will be enrolled. The outcome assessor will be blind to the group assignment of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- target of Stroke Volume Variation ≤ 6% (Experimental): The rate of intraoperative fluid administration will be adjusted to achieve the target of Stroke Volume Variation ≤ 6%. A crystalloid bolus of 200 ml will be repeatedly administered every 20 min until the target was achieved. The basal rate of fluid administration will be 3 ml/kg/hr.
  Interventions: Other: Crystalloid fluid administration with the target of stroke volume variation ≤ 6%
- target of Stroke Volume Variation ≤ 12% (Active Comparator): The rate of intraoperative fluid administration will be adjusted to achieve the target of Stroke Volume Variation ≤ 12%. A crystalloid bolus of 200 ml will be repeatedly administered every 20 min until the target was achieved. The basal rate of fluid administration will be 3 ml/kg/hr.
  Interventions: Other: Crystalloid fluid administration with the target of stroke volume variation ≤ 12%

INTERVENTIONS:
Other: Crystalloid fluid administration with the target of stroke volume variation ≤ 12% — The rate of crystalloid fluid administration will be controlled to achieve the target of stroke volume variation ≤ 12%
  Arms: target of Stroke Volume Variation ≤ 12%
Other: Crystalloid fluid administration with the target of stroke volume variation ≤ 6% — The rate of crystalloid fluid administration will be controlled to achieve the target of stroke volume variation ≤ 6%
  Arms: target of Stroke Volume Variation ≤ 6%

SUMMARY:
The investigators sought to compare the effect of two preload targets of stroke volume variation of ≤6% and ≤12% on the postoperative renal function in patients undergoing living donor kidney transplantation. Goal-directed fluid therapy will be performed in both groups to maintain adequate stroke volume, stroke volume variation, mean arterial pressure (or systemic vascular resistance) during kidney transplantation. Only the preload target for giving crystalloid during surgery will be different between groups.

DETAILED DESCRIPTION:
The adequate preload target of fluid management has not yet been established during kidney transplantation. Traditionally, sufficient intravascular volume status has been recommended to maintain perfusion to renal graft. Stroke volume variation was reported to be superior to the traditional target of central venous pressure. In this regard, the investigators sought to compare the effect of two preload targets of stroke volume variation of ≤6% and ≤12% on the postoperative renal function in patients undergoing living donor kidney transplantation. Goal-directed fluid therapy will be performed in both groups to maintain adequate stroke volume, stroke volume variation, mean arterial pressure (or systemic vascular resistance) during kidney transplantation. Only the preload target for giving crystalloid during surgery will be different between groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients who are undergoing living donor kidney transplantation with continuous radial artery pressure monitoring

Exclusion Criteria:

* Patients who have cardiac arrhythmia of atrial fibrillation, multiple ventricular premature complex
* Cardiac systolic dysfunction with left ventricle ejection fraction <50%
* Continuous arterial pressure monitoring at the site other than radial artery.
* Patients who are considered to be intolerant to rapid fluid administration

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
serum neutrophil-gelatinase-associated lipocalin (NGAL) | at the end of surgery
  urine biomarker of renal injury

SECONDARY OUTCOMES:
serum neutrophil-gelatinase-associated lipocalin (NGAL) | at the anesthesia induction procedure
  urine biomarker of renal injury
Delayed graft function determined by the incidence of hemodialysis | during the first postoperative week
  Delayed graft function determined by the incidence of hemodialysis
Delayed graft function determined by urine output (less than 1200 ml) | during the first postoperative day
  Delayed graft function determined by urine output (less than 1200 ml)
Delayed graft function determined by serum creatinine | during the 48 hours after surgery
  Delayed graft function determined by serum creatinine (No decrease in creatinine of more than 10% of preoperative value)
Delayed graft function determined by serum creatinine (more than 2.5 mg/dL) | during the 10 days after surgery
  Delayed graft function determined by serum creatinine (more than 2.5 mg/dL)
Delayed graft function determined by glomerular filtration rate | during the 24 hours after surgery
  Delayed graft function determined by glomerular filtration rate (less than 10 ml/min/m2)
Delayed graft function determined by serum creatinine (do not decrease less than preoperative value) | during the first postoperative week
  Delayed graft function determined by serum creatinine (do not decrease less than preoperative value)
Immediate graft function | after eight days after surgery
  serum creatinine decrease less than 70% of preoperative value
slow graft function | after eight days after surgery
  serum creatinine decrease greater than 70% of preoperative value
serum creatinine value | first postoperative day
  serum creatinine value
serum creatinine value | third postoperative day
  serum creatinine value
serum creatinine value | seventh postoperative day
  serum creatinine value
Incidence of pneumonia | during the first postoperative week
  Incidence of pneumonia
Incidence of wound infection | during the first postoperative week
  Incidence of wound infection
Incidence of postoperative bleeding | during the first postoperative week
  Incidence of postoperative bleeding
hospital length of stay | the first postoperative month
  hospital length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No